CLINICAL TRIAL: NCT01435343
Title: Multicenter, Prospective, Open-label, Single-arm, Phase I-II Clinical Trial to Analyze Induction Therapy With a Combination of Fludarabine, Idarubicin, Cytarabine, G-CSF and Plerixafor for the Treatment of Young Patients With Relapsed or Refractory AML
Brief Title: Treatment of Relapsed or Refractory Acute Myeloblastic Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLERIFLAG
Record Dates: First submitted 2011-09-14; First posted 2011-09-16 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2016-09

CONDITIONS: Acute Myeloblastic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — fludarabine; Idarubicin; Cytarabine; Granulocyte Colony-Stimulating Factor; plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: fludarabine — 30 mg/m2/day intravenously on days 1 to 4
Drug: Idarubicin — 10 mg/m2/day intravenously on days 1 to 3
Drug: cytarabine — 2 g/m2/day intravenously on days 1 to 4
Drug: G-CSF — 5 μg/kg/day subcutaneously from days 1 to 4
Drug: plerixafor — intravenously from days 1 to 4

SUMMARY:
Second-line induction therapy with fludarabine, idarubicin, cytarabine,Granulocyte colony-stimulating factor (G-CSF) and plerixafor, in patients with relapsed or refractory Acute Myeloblastic Leukemia (AML) aged 65 or younger.

DETAILED DESCRIPTION:
This protocol corresponds to a multicenter, open-label, non-randomized, Phase I-II study designed to determine the safety and efficacy of the combination of plerixafor with chemotherapy in young patients with relapsed or refractory AML.

The clinical trial is divided into pre-treatment and treatment periods (induction and consolidation cycle(s) and consists of two general phases: an initial Phase I in which escalating doses of plerixafor will be given to 4 groups, each with 3 patients; and a secondary Phase II in which an additional patient group will be treated with the maximum tolerated dose (MTD) from Phase I.

In the pre-treatment period, all patients who provide written informed consent will be screened and any patients who meet all the inclusion and none of the exclusion criteria will be eligible for treatment.

The patients who are finally included in the study should begin treatment within 7 days after signing the informed consent document (ICD). The pre-treatment period begins when the ICD is signed and enrollment occurs when the patient receives the first study drug of the treatment regimen (i.e., Day 1 of the induction cycle).

In this study, the induction cycle will consist of fludarabine 30 mg/m2/day intravenously on days 1 to 4, idarubicin 10 mg/m2/day intravenously on days 1 to 3, cytarabine 2 g/m2/day intravenously on days 1 to 4, G-CSF 5 μg/kg/day subcutaneously from days 1 to 4, and plerixafor intravenously from days 1 to 4. The dose of plerixafor will be escalated over 4 groups of three patients as follows: 240 μg/kg/day (120 μg/kg/12 h); 320 μg/kg/day (160 μg/kg/12 h); 400 μg/kg/day (200 μg/kg/12 h); and 480 μg/kg/day (240 μg/kg/12 h). If MTD is observed with the first treatment dose of plerixafor the dose will be progressively deescalated to 160 μg/kg/day (80μg/kg/12 h) on a first deescalating level or 240 μg/kg/day in a single daily dose on a second deescalating level if no twice a day (BID) dose is tolerated. Patient enrollment will be expanded to a total of 55 patients using MTD. If patients do not achieve CR after one induction cycle they will leave the study and be followed according to routine clinical practice. Patients who achieve complete response (CR) who are eligible for allogeneic hematopoietic stem cell transplantation (HSCT) and have a donor will leave the trial and receive allogeneic HSCT and will be followed according to routine clinical practice. Patients who achieve CR and are not eligible for allogeneic HSCT or do not have a donor will receive two consolidations with cytarabine at 3 g/m2/12 hours on days 1, 3 and 5 along with Granulocyte colony-stimulating factor (GCSF) at 5 μg/kg/day on days 1 to 5 and plerixafor at the same dose used in the induction cycle on days 1, 3 and 5, coinciding with the days that cytarabine is administered.

In the context of this protocol, a treatment cycle is defined as the first day of the study drug administration regimens (Day 1) up to and including the day before the first day of the treatment cycle immediately afterwards. The treatment cycles will begin after Day 28 but no later than Day 85, counting from Day 1 of the treatment cycle immediately before.

Patients will be assessed in the three days before each cycle (see Appendix A). Follow-up, outside the protocol in routine clinical practice, will be performed monthly during the first year and at least every three months during the second year; notwithstanding, visits may be more frequent at the discretion of each site or based on the clinical characteristics.

All treatment cycles will be administered while the patient is hospitalized. Clinical procedures for the care of patients with acute leukemia require flexibility. However, deviations from the study treatment defined in this section must be prospectively discussed with the coordinator.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AML according to the WHO criteria
* Relapsed or refractory AML as defined below First relapse after standard treatment with duration of the first remission less than year
* Refractoriness to an induction cycle that includes cytarabine and anthracyclines
* Nonpromyelocytic leukemia (absence of t(15;17) or PML-RARα rearrangement and its variants)
* Peripheral blood blast cell count less than 50 x 109/L. Hydroxyurea and leukopheresis can be used to lower the blast count prior to beginning treatment
* Age ≤ 65 years and ≥ 18 years
* ECOG performance status of 0-2
* Provide signed written informed consent
* Be able to comply with study procedures and follow-up examinations
* Be nonfertile or agree to use birth control during the study through the end of last treatment visit
* Adequate renal and hepatic function as indicated by all of the following:

Total bilirubin <1.5 x Institutional Upper Limit of Normal (ULN); and AST and ALT <2.5 xULN; and Serum creatinine <1.0 mg/dL; if serum creatinine <1.0 mg/dL, then, the estimated glomerular filtration rate (GFR) must be <60 ml/min/1.73 m2 as calculated by the Modification of Diet in Renal Disease (MDRD) equation - Minimal impairment of cardiac function as measured by at least 1 of the following: Left ventricular ejection fraction (LVEF) >40% on multigated acquisition (MUGA) scan or radionuclide angiographic scan; or Left ventricular fractional shortening >22% on echocardiography exam;

Exclusion Criteria:

* Diagnosis of acute promyelocytic leukemia (APL, French-American-British [FAB] classification M3 or WHO classification of APL with t(15;17)(q22;q12), (PML/RARalfa and variants)
* AML secondary to previous treatment for myelodysplastic syndrome (MDS)
* Peripheral blood blast cell count ≥ 50 x 109/L. Hydroxyurea and leukopheresis can be used to lower the blast count prior to beginning treatment
* Prior investigational treatment within 30 days prior to the first dose of study drug. If any investigational treatment has been received prior to this time point, drug related toxicities must have recovered to Grade 1 or less prior to first dose of study drug
* Prior hematopoietic stem cell transplant (HSCT) (previous autologous hematopoietic stem cell transplant is allowed)
* Investigational agent received within 5 days prior to the first dose of study drug. If received any investigational agent prior to this time point, drug-related toxicities must have recovered to Grade 1 or less prior to first dose of study drug
* Impaired renal and liver function as indicated by the following:

Total bilirubin > 1.5 x upper limit of normal (ULN) provided that this is not attributable to AML itself; or AST and ALT > 2.5 xULN provided that this is not attributable to AML itself; or Serum creatinine > 1.0 mg/dL provided that the estimated glomerular filtration rate (GFR) is ≤ 60 mL/min/1.73 m2 as calculated by the Modification of Diet in Renal Disease (MDRD) equation

- Impaired cardiac function as measured by at least 1 of the following: Left ventricular ejection fraction (LVEF) < 40% on multigated acquisition (MUGA) scan or radionuclide angiographic scan; or Left ventricular fractional shortening < 22% on echocardiography exam;

* Poor overall condition ECOG 3-4
* Refusal to sign the informed consent
* Unable to comply with study procedures and follow-up examinations
* Psychiatric disorders that could interfere with consent, study participation or follow-up
* Systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment)
* Diagnosis of another malignancy, unless the patient has been disease-free for at least 5 years following the completion of curative intent therapy with the following exceptions:

Patients with treated non-melanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia, regardless of the disease-free duration, are eligible for this study if definitive treatment for the condition has been completed Patients with organ-confined prostate cancer with no evidence of recurrent or progressive disease based on prostate-specific antigen (PSA) values are also eligible for this study if hormonal therapy has been initiated or a radical prostatectomy has been performed

* Clinical evidence suggestive of central nervous system (CNS) involvement with leukemia unless a lumbar puncture confirms the absence of leukemic blasts in the cerebrospinal fluid (CSF)
* Prior positive test for the human immunodeficiency virus (HIV)
* History of hypersensitivity to any of the study drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2012-07; Primary Completion 2016-05 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Efficacy in terms of number of complete responses | 1 year

SECONDARY OUTCOMES:
Safety in terms of percentages of adverse events presented | 1 year

CONTACTS AND LOCATIONS:
Locations (10):
- Spain (10):
  - Hospital Universitari Germans Trials i Pujol, Badalona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau., Barcelona
  - Hospital Duran i Reynals - ICO L'Hospitalet, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Hospital Universitari La Fe, Valencia

REFERENCES:
- [Derived] Martinez-Cuadron D, Boluda B, Martinez P, Bergua J, Rodriguez-Veiga R, Esteve J, Vives S, Serrano J, Vidriales B, Salamero O, Cordon L, Sempere A, Jimenez-Ubieto A, Prieto-Delgado J, Diaz-Beya M, Garrido A, Benavente C, Perez-Simon JA, Moscardo F, Sanz MA, Montesinos P; CETLAM and PETHEMA groups. A phase I-II study of plerixafor in combination with fludarabine, idarubicin, cytarabine, and G-CSF (PLERIFLAG regimen) for the treatment of patients with the first early-relapsed or refractory acute myeloid leukemia. Ann Hematol. 2018 May;97(5):763-772. doi: 10.1007/s00277-018-3229-5. Epub 2018 Feb 2. PMID 29392425
- See also: CRO — http://www.cabyc.com